CLINICAL TRIAL: NCT04455659
Title: Impact of Adding Transcutaneous Electrical Nerve Stimulation to Conventional Physical Therapy Exercise on Pain Relief Among Patients With Pudendal Neuralgia.
Brief Title: Impact of Adding TENS to Conventional Physical Therapy Exercise on Pain Relief Among Patients With Pudendal Neuralgia.
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Lecturer , department of physical therapy for surgery, Faculty of Physical Therapy , Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1720
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Pudendal Neuralgia
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS + Conventional physical therapy exercise (Experimental)
  Interventions: Device: Trans-cutaneous Electrical Nerve Stimulation; Procedure: Conventional physical therapy exercise
- conventional physical therapy exercise (Active Comparator)
  Interventions: Procedure: Conventional physical therapy exercise

INTERVENTIONS:
Device: Trans-cutaneous Electrical Nerve Stimulation — TENS that was applied once daily, three times per week for 8 weeks. Each treatment session was conducted for 20 minutes, two electrodes were positioned over the perineal area between anus and scrotum on the Centrum tendineum, while the other two electrodes were applied under the buttocks medially at the level of the ischial spines (medial to the ischial spines bilaterally) with the patient in comfortable supine hook-lying position with abducted hips. to prevent burn beneath the electrodes, the surface area of the electrode should be equal to or greater than 4 cm2 to minimize the heat production. In addition, to decrease the current density between electrodes, the inter-electrode distance was less than the cross sectional area of the electrode
  Other Names: Conventional physical therapy exercise
  Arms: TENS + Conventional physical therapy exercise
Procedure: Conventional physical therapy exercise — physical therapy program for 30 minutes, and 3 times per week for 8 weeks in the form of strengthening exercise, clam - shell exercise, and stretching exercise focusing on obturator internus muscle, range of motion exercise for the hip and pelvis musculature for 30 minute three times a week for consecutive 8 weeks , each type of exercise was performed for a duration of 6 seconds and repeated 10 times

SUMMARY:
Fifty two male participants, 30-50 years old, suffering from chronic pudendal neuralgia were randomly assigned either into experimental group (26 patients) received TENS plus the traditional physical therapy program( including range of motion exercise, stretching exercise of obturator internus muscle, clam shell exercise, relaxation exercise and underwater exercise) 3 sessions per week for 8 successive weeks, or control group (26 patients) received only the traditional physical therapy exercise for the same period of time. Intensity of pain by Verbal rating scale (VRS) as well as Serum cortisol level (SCL)and Etodolac level intake are measured pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male with ages ranged from 30 to 50 years.
* Suffering from pudendal neuralgia and its intractable perineal pain that persists for a minimum one month beyond the acute onset.
* Pelvic pain with sitting that relived by standing or toilet sitting.
* Anal pain, dyspareunia and genital pain

Exclusion Criteria:

* Those who had history of skin malignancy.
* Diabetic,
* Sensory disorders,
* Circulatory insufficiency
* Acute infection of the treatment area,
* Renal failure

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Pain intensity (NRS) | 8 weeks of treatment
  Numeric Rating Scale (NRS) for pain is a one-dimensional measure of pain intensity in adults, including those with chronic pain .It is an instrument tool to measure the intensity of pain, Numerical pain rating scale consists an 11-point numeric scale with 0 representing "no pain" and 10 representing extreme pain (Worst possible pain)

SECONDARY OUTCOMES:
Serum cortisol level | 8 weeks of treatment
  A venous blood sample of 8 CC was taken at the morning, centrifuged and stored at 20ºC till analyzed, Normal cortisol level ranged from 9-25 µg/dL at morning and patients with painful conditions tended to have higher than normal SCL
Calculation of Etodolac Intake (ELI) in mg | 8 weeks of treatment
  It was done before and after the treatment program

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we will share study protocol after 6 months from publication.
Supporting Information: Study Protocol, ICF
Time Frame: After 6 months from publication.